CLINICAL TRIAL: NCT05055934
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase II Dose Exploratory Study to Evaluate the Effectiveness and Safety of SHR-1314 Injection in Adult Subjects With Active Psoriatic Arthritis
Brief Title: Study of the Effectiveness and Safety of SHR-1314 for Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1314-204
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2021-09

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1314 injection (Experimental)
  Interventions: Drug: SHR-1314 injection
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SHR-1314 injection — SHR-1314 injection
  Arms: SHR-1314 injection
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This study is a randomized, double-blind, multicenter, placebo-controlled Phase II clinical study, consisting of a 4-week screening period, a 12-week core treatment period, a 12-week maintenance treatment period, and an 8-week safety follow-up period. It is planned to include 111 adult subjects with psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily signs an informed consent form before any procedures related to the research start;
2. Age ≥18 years old and ≤75 years old at the time of signing the informed consent form, regardless of gender;
3. At the time of screening, it met the 2006 psoriatic arthritis classification standard (CASPAR);
4. There is active PsA before randomization;
5. Have active plaque psoriasis (at least one plaque skin lesion) at the time of screening, or have a history of plaque psoriasis;

Exclusion Criteria:

1. Existence of any of the following medical history or comorbid diseases: drug-induced psoriasis; other active inflammatory diseases or autoimmune diseases; history of organ transplantation; history of lymphocytic proliferation; severe infections, etc.
2. Have received psoriatic arthritis or psoriasis drugs, such as intra-articular injections, plant preparations, etc. within a certain period of time in the past.
3. Those who are allergic to the drug ingredients or excipients in this study, or are allergic to other biological agents.
4. A history of alcohol abuse or illegal drug abuse in pregnant or breastfeeding women, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving ACR 20 improvement at week 12 | at week 12

SECONDARY OUTCOMES:
The proportion of subjects who achieved ACR 50 improvement (week 12) | week 12
The proportion of subjects who achieved ACR 70 improvement (week 12) | week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital of the Shanghai FuDan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xue Y, Sun L, Zhang N, Chen H, Shi X, Liu S, Chen L, Ma X, Wei H, Jiang Z, Li X, Fan H, Li H, Li J, Wu R, Shi G, Zhu J, Kong X, Lu Y, Liu P, Zheng Q, Bai X, Zhang S, Wan W, Zou H. Vunakizumab in patients with active psoriatic arthritis: a multicentre, randomized, double-blind, placebo-controlled, phase 2 study. Rheumatology (Oxford). 2026 Feb 3:keag060. doi: 10.1093/rheumatology/keag060. Online ahead of print. PMID 41632483